CLINICAL TRIAL: NCT00287222
Title: Bevacizumab and Erlotinib in Inoperable and Metastatic Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Rangaswamy Govindarajan, UAMS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UARK 2005-13
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Inoperable and Metastatic Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 - Bevacizumab/Erlotinib (Experimental): Subjects will be treated with bevacizumab and erlotinib
  Interventions: Drug: Bevacizumab; Drug: Erlotinib

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/KG I.V. every 21 days
  Other Names: Avastin
Drug: Erlotinib — 150 mg orally every day
  Other Names: Tarceva

SUMMARY:
The primary efficacy endpoint will be the proportion of subjects that remain free of progression at the 27th week following the onset of treatment. Secondary objectives include the subject's time in weeks from treatment onset to documented disease progression as assessed by the RECIST criteria, response rate, median and overall survival, safety and tolerability.

DETAILED DESCRIPTION:
This is a phase II study to assess the proportion of subjects that remain progression-free by the 27th week following the onset of treatment and to assess the efficacy of the combination of Bevacizumab and Erlotinib in prolonging time to progression in subjects with inoperable and metastatic hepatocellular carcinoma. Subjects will be treated with a combination of rhuMAb VEGF (Bevacizumab), in combination with Erlotinib and TTP will be assessed as per RECIST criteria. The disease will be evaluated at base line and every 9 weeks with CT scan/MRI and AFP levels. Subjects will be kept on the study till disease progression (as defined by RECIST criteria) or death.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have histologically or cytologically confirmed diagnosis of hepatocellular carcinoma, regardless of biopsy site.
* Subjects with a liver mass and markedly elevated AFP (>500ng/mL) are eligible.
* Subjects should not be on the liver transplantation schedule
* Subjects can have prior therapy with sorafenib (nexavar) only if the therapy was stopped due to toxicity or allergic reaction soon after starting. Subjects must have been treated for less than two weeks to be eligible.
* Radiation therapy for palliation to the areas outside the site of tumor used for measurements is permitted. If a subject has received radiation therapy to the liver, the subject id eligible if there is a new lesion or if the prior lesion has increased in size.
* Subjects who have recovered from prior surgical procedure
* Performance status of ECOG 0-2
* Measurable or evaluable disease
* Be declared unresectable or not suitable candidates for surgery
* Adequate organ functions
* Serum bilirubin <3 mg/dl, AST <5x ULN, ALT <5XULN
* Serum albumin >2.5 g/dl
* Serum creatinine < 2.0 mg/dl
* ANC >1200 MM3
* Platelet count >75,000/ml
* PT/INR < 1.5 X ULN
* Life expectancy of >3 months
* Subjects should be able to sign informed consent and be agreeing to comply with therapy and follow up.
* Negative pregnancy test in women with childbearing potential, within one week prior to initiation of treatment.
* Fertile men and women must agree to use adequate contraception prior to study entry, for the duration of study participation, and for at least 1 week after therapy.
* Age >/= 18 years. The agents Bevacizumab and Erlotinib have not been studied in pediatric subjects, thus the doses to be used in this study cannot be assumed to be safe in children.

Exclusion Criteria:

* Surgically resectable disease
* Subjects with active bacterial infections
* Subjects with brain metastases
* Pregnant women (positive pregnancy test) or lactating
* No other malignancy is allowed except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer or other cancer for which the subject has been disease-free for five years.
* Abnormalities of the cornea based on history (e.g. dry eye syndrome, Sjogren's syndrome) or congenital abnormality (e.g. Fuch's dystrophy).
* Current, recent (within 4 weeks of the first infusion of the study), or planned participation in an experimental drug study other than a Genentech-sponsored Bevacizumab/Erlotinib cancer study
* Hepatic encephelopathy (as per treating physician's evaluation)
* Uncontrolled blood Pressure >150/100 mmHg
* Unstable angina
* NYHA grade II or greater congestive heart failure
* History or myocardial infraction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease (clinically significant venous or arterial thrombotic disease).
* Evidence of bleeding diathesis or coagulopathy
* Urine protein: creatinine ratio >1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to comply with study and/or follow-up procedures
* Gastrointestinal disease resulting in an inability to take oral medication or a requirement for intravenous hyperalimentation.
* History of significant gastrointestinal bleeding requiring procedural intervention (e.g. variceal banding, TIPS procedure, arterial embolization, topical coagulation therapy) within six months prior to study Day 0.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rangaswamy Govindarajan, MD, Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kansas University Medical Center, Kansas City, Kansas

REFERENCES:
- [Derived] Govindarajan R, Siegel E, Makhoul I, Williamson S. Bevacizumab and erlotinib in previously untreated inoperable and metastatic hepatocellular carcinoma. Am J Clin Oncol. 2013 Jun;36(3):254-7. doi: 10.1097/COC.0b013e318248d83f. PMID 22643560

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period was from 7/08/2005 to 12/17/2008. Recruitment occurred at the University of Arkansas for Medical Sciences medical oncology clinic and Kansas University Cancer Center.
Groups:
- Bevacizumab and Erlotinib: Subjects will be treated with bevacizumab and erlotinib
Period: Overall Study
Arm/Group | Bevacizumab and Erlotinib
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and Erlotinib
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Remained Free of Progression at the 27th Week.
Time Frame: 27 weeks
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Bevacizumab and Erlotinib
Number analyzed (Participants) | 21
participants | 21
Statistical Analysis 1: Comparison: Bevacizumab and Erlotinib; Estimating the percentage of participants that remain free of disease progression at 27 weeks from the onset of treatment, and testing that proportion against a null-hypothesis proportion of 0.04 using the one-sided exact binomial test at 5% alpha, based upon historical data from the literature; Test type: Superiority or Other; p = 0.0006, one-sided exact binomial test; percentage progression free at 27 weeks = 28, 95% CI 2-sided [10 to 53], Standard Error of Mean 10.97

ADVERSE EVENTS:
Arm/Group | Bevacizumab and Erlotinib
Serious Adverse Events (participants affected / at risk) | 11/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and Erlotinib (N=21)
Fatigue (General disorders) | 4 (4)
dehydration (Metabolism and nutrition disorders) | 2 (2)
hematemesis (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Two subjects withdrew consent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No